CLINICAL TRIAL: NCT05523232
Title: Effects of Localized Vibration Training on the Biceps Brachii Muscle and Grip Strength in Healthy Adult Males: An Experimental Study
Brief Title: Effects of Vibrations on the Biceps Brachii Muscle and Grip Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RRC-2018-003
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Muscle Strength
Keywords: Vibration Training; Biceps Brachii; Muscle Strength; Handgrip

STUDY DESIGN:
Intervention Model Description: Two group parallel design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 42 Hz group (Experimental): Vibration training with 42 Hz was given to participants.
  Interventions: Other: Vibration training with 42 Hz
- 63 Hz group (Active Comparator): Vibration training with 63 Hz was given to participants.
  Interventions: Other: Vibration training with 63 Hz

INTERVENTIONS:
Other: Vibration training with 42 Hz — Vibration exposure was given using a handheld vibration device.
  Arms: 42 Hz group
Other: Vibration training with 63 Hz — Vibration exposure was given using a handheld vibration device.
  Arms: 63 Hz group

SUMMARY:
It has been suggested that applying acute vibration exercises enhances muscle force, like several weeks of resistance training. The present study investigated the effects of local vibration with two different frequencies on biceps brachii isometric muscle strength and grip strength in healthy young men. Isometric strength of the biceps brachii muscle and grip strength were assessed at baseline and after vibration training (immediate, 10 minutes, and 20 minutes post vibration training).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males

Exclusion Criteria:

* history of recent upper extremity injury
* sensory deficits in the upper extremity
* history of recent upper extremity surgery
* participation in any resistance training

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Isometric strength of Biceps brachii muscle | 20 minutes
  Isomeric strength of the biceps brachii muscle of the dominant arm was measured at an Angle of 90 degree flexion using a handheld dynamometer
Hand grip strength | 20 minutes
  Hand grip strength was measured using a standard adjustable Jamar hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No